CLINICAL TRIAL: NCT02145130
Title: A Phase I, Two Armed, Open, Prospective and Multicentre Study to Evaluate the Safety of Autologous Tissue-engineered Dermal Substitutes and Dermo-epidermal Skin Substitutes for the Treatment of Large Deep Partial and Full Thickness Skin Defects in Children and Adults
Brief Title: Phase I Study for Autologous Dermal Substitutes and Dermo-epidermal Skin Substitutes for Treatment of Skin Defects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University Hospital, Zürich (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EuroSkinGraft / ESG-01-2011
Record Dates: First submitted 2014-05-20; First posted 2014-05-22 (Estimated); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Burn Injury; Soft Tissue Injury; Skin Necrosis; Scars; Congenital Giant Nevus; Skin Tumors
Keywords: Skin; Tissue-engineering; Autologous; Dermis; Epidermis
MeSH Terms: conditions — Burns; Soft Tissue Injuries; Necrosis; Cicatrix; Skin Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- denovoDerm (Experimental): Autologous tissue-engineered dermal substitute
  Interventions: Biological: denovoDerm
- denovoSkin (Experimental): Autologous tissue-engineered dermo-epidermal skin substitute
  Interventions: Biological: denovoSkin

INTERVENTIONS:
Biological: denovoDerm — Transplantation of an autologous tissue-engineered dermal substitute, covered with autologous split-thickness skin
  Arms: denovoDerm
Biological: denovoSkin — Transplantation of autologous tissue-engineered dermo-epidermal skin substitute, no additional coverage needed
  Arms: denovoSkin

SUMMARY:
The purpose of this study is the evaluation of the safety of autologous tissue-engineered dermal substitutes "denovoDerm" (first arm) and dermo-epidermal skin substitutes "denovoSkin" (second arm) transplanted onto the wound bed in children and adults.

ELIGIBILITY:
Inclusion Criteria:

* Deep partial or full thickness skin defect of at least 9 cm2 requiring surgical wound coverage due to:

  1. Acute cases: burn injury, soft tissue injury, skin necrosis after purpura fulminans
  2. Reconstructive cases (elective surgery): scar formation after burn injuries, congenital giant nevus, skin tumours
* Informed consent by patients/parents or other legal representatives

Exclusion Criteria:

* Infected wounds or positive general microbiological swabs taken from the nose for multi-resistant germs
* Patients tested positive for HBV, HCV, syphilis or HIV
* Patients with known underlying or concomitant medical conditions that may interfere with normal wound healing (e.g. immune deficiency, systemic skin diseases, any kind of congenital defect of metabolism including diabetes)
* Coagulation disorders as defined by INR outside its normal value, PTT >ULN and fibrinogen <LLN and / or at the Investigator's discretion
* Previous enrolment of the patient into the current study
* Participation of the patient in another study within 30 days preceding and during the present study
* Patients or parents/other legal representatives expected not to comply with the study protocol
* Suspicion of child abuse
* Pregnant or breast feeding females
* Contamination derived from biopsy which could interfere with patients health
* Due to patient derived variations, isolated cells from biopsy do not proliferate or proliferate insufficiently
* Skin substitute has not been released due to production specific deviations
* Patients allergic to amphotericin B and gentamicin

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-05; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Safety | denovoDerm: 4-6 days and 21 days after transplantation, denovoSkin 9-11 days and 21 days after transplantation
  Assessment/reporting of local infection rate and graft take

SECONDARY OUTCOMES:
Adverse events | until 90 days post transplantation
  Assessment/reporting of number of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Böttcher, PD Dr. med., Principal Investigator — University Children's Hospital, Zurich
Locations (2):
- Switzerland (2):
  - University Children's Hospital Zurich: denovoDerm, Zurich, Canton of Zurich
  - University Children's Hospital Zurich: denovoSkin, Zurich, Canton of Zurich

REFERENCES:
- [Derived] Schiestl C, Neuhaus K, Meuli M, Farkas M, Hartmann-Fritsch F, Elrod J, Bressan J, Reichmann E, Bottcher-Haberzeth S. Long-Term Outcomes of a Cultured Autologous Dermo-Epidermal Skin Substitute in Children: 5-Year Results of a Phase I Clinical Trial. J Burn Care Res. 2025 Mar 4;46(2):326-334. doi: 10.1093/jbcr/irae150. PMID 39115183